CLINICAL TRIAL: NCT01953679
Title: A Phase IIb Randomized, Double Blind, Comparative Study to Assess the Efficacy, Safety, Tolerability and Inhibition of Ovulation of Two Continuous Regimens of Oral Daily 5 mg or 10 mg of Ulipristal Acetate (UPA), Versus a Dose of 5.0mg UPA for 24/4 Days
Brief Title: Efficacy Study of Two Continuous Regimens of Oral Daily 5 mg or 10 mg of Ulipristal Acetate (UPA), Versus a Dose of 5.0mg UPA for 24/4 Days
Acronym: CCN013
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Premier Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CCN013
Record Dates: First submitted 2013-08-23; First posted 2013-10-01 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Focus: Estrogen-free Oral Contraception
MeSH Terms: interventions — ulipristal acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5mg UPA (Active Comparator): Continuous regimen of oral daily 5 mg of ulipristal acetate (UPA) versus a cyclic regimen of 5 mg UPA for 24 days followed by a 4 day hormone free interval.
  Interventions: Drug: Ulipristal Acetate
- 10mg UPA (Active Comparator): Continuous regimen of oral daily 10 mg of ulipristal acetate (UPA) versus a cyclic regimen of 5 mg UPA for 24 days followed by a 4 day hormone free interval.
  Interventions: Drug: Ulipristal Acetate

INTERVENTIONS:
Drug: Ulipristal Acetate

SUMMARY:
To compare the pharmacodynamic effects of 2 continuous dose regimens of ulipristal acetate 5.0 and 10.0 mg-only oral contraception, versus a 24/4 day regimen of UPA 5.0 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 18 and 35 years old.
2. In good health, with regular menstrual cycles that occur every 21-35 days.

   1. If subject is postpartum or post-abortal (with abortion in second trimester), she will be required to have two normal menstrual cycles (3 menses) prior to screening.
   2. If subject had an abortion in the first trimester, she will be required to have at least one menstrual cycle (two menses) prior to screening.
3. No current use of hormonal contraception or an intrauterine device and having had at least one complete menstrual cycle since having stopped hormonal contraception before starting the treatment.

   a. No use of injectable contraceptives (e.g. cyclofem or depo-medroxyprogesterone acetate) during the 6 months prior to screening unless the subject has returned to normal menses since last injection.
4. Have a negative urine pregnancy test at the admission visit.
5. Will not be at risk for pregnancy. They will be consistently using a non-hormonal method, barrier method with every act of intercourse until the time of study exit OR have a surgically sterile male partner with a vasectomy, must have undergone previous tubal ligation, be abstinent, or be in a same-sex relationship from the control period through study exit (including recovery period).
6. In the opinion of the investigator, willing and able to follow all study requirements, including use of the study product and willing to record requested information on a daily diary.
7. Understand and sign an IRB approved inform consent form prior to screening activities (including fasting blood draws).
8. Will have diastolic blood pressure (BP) ≤95 mm Hg and systolic BP ≤145 mm Hg after 5 minutes in sitting position.
9. BMI < 40 kg/m2 and not having previously undergone bariatric surgery.
10. Agree not to participate in any other clinical trials during the course of this study.

Exclusion Criteria:

1. Women less than 18 and older than 35 years old.
2. Women with menstrual cycle length of less than 21 or more than 35 days; or with spontaneous irregular menstrual cycle length with intra-individual variations of more than 5 days.

   a. If subject is postpartum or post-abortal (with abortion in second trimester) and not had two normal menstrual cycles (3 menses) prior to screening.

   b. If subject had an abortion in the first trimester and not had at least one menstrual cycle (two menses) prior to screening.
3. Currently pregnant as confirmed by positive high-sensitivity urine pregnancy test.
4. Unwilling to use a barrier method with every act of intercourse until study exit OR not have a surgically sterile male partner with a vasectomy, not have undergone previous tubal ligation, not abstinent, or not in a same-sex relationship from the control period through study exit (including recovery period).
5. Women planning pregnancy within their months of study participation.
6. Currently breast-feeding or within 30 days of discontinuing breast feeding, unless the woman has already had a menses following discontinuation of breast feeding.
7. Current use of an IUD, or other hormonal contraception within last complete menstrual cycle prior to screening.

   a. Use of injectable contraceptives (e.g. cyclofem or depo-medroxyprogesterone acetate) during the 6 months prior to screening without the subject returning to normal menses since last injection.
8. Undiagnosed abnormal genital bleeding.
9. Known hypersensitivity to the active substance UPA or any of the excipients of the study treatment.
10. Anomalies in endometrial appearance, TVUS or safety labs done at screening visit recognized as clinically significant by the investigator.
11. Subject with a previous history of endometrial ablation.
12. A clinically significant Pap test abnormality, as managed by current local or national guidelines. Women with a current abnormal Pap (within the last eighteen months):

    1. In accordance with the Bethesda system of classification: smear suggestive of high-grade pre-cancerous lesion(s), including high grade squamous intraepithelial lesions (HGSILs), are excluded; • Women with low grade squamous intraepithelial lesion (LGSIL) or atypical squamous cells of undetermined significance (ASCUS)/high-risk human papillomavirus (HPV) positive, or Atypical squamous cells, cannot rule out a high grade lesion (ASC-H) may participate if further evaluated with colposcopy and biopsy determines no evidence of a lesion with a severity greater than cervical intraepithelial neoplasia (CIN) I. • Women with a biopsy finding of CIN I should have follow-up for this finding per standard of care; women are excluded if treatment is indicated.
    2. In accordance with other Pap class systems:

       • Women with high grade dysplasia are excluded.

       • Women with atypical glandular cells of undetermined significance (AGUS) are excluded.

       • Women with low grade dysplasia or CIN I interpretation on Pap test may participate following exclusion of a high grade lesion by colposcopic evaluation based on Investigator discretion and provided there is appropriate follow up in accordance with local standards.
13. Has any of the following known contraindication to progestin-only oral contraceptive (OC):

    1. History or existing breast cancer, or other hormone sensitive neoplasia;
    2. Current and history of ischemic heart disease or stroke while pregnant or taking birth control pills;
    3. Acute deep venous thrombosis or pulmonary embolism;
    4. Systemic Lupus Erythematosus with positive or unknown antiphospholipid antibodies;
    5. Benign and malignant liver tumors;
    6. Severe (decompensated) cirrhosis.
14. Hereditary galactose intolerance, Lapp lactase deficiency , or glucose-galactose malabsorption.
15. Known or suspected alcoholism or drug abuse.
16. Known HIV infection.
17. Smoking 15 cigarettes or more per day must be evaluated by the investigator or medically qualified designee for inclusion based on risk factors that would increase their risk for cardiovascular disease (CVD) and thromboembolism.
18. Current or past deep vein thrombophlebitis or thromboembolic disorders.
19. Current or past medically diagnosed severe depression, which, in the opinion of the investigator, could be exacerbated by use of a hormonal contraceptive, unless she is stable on antidepressant medication.
20. Concomitant use of medication thought to interact with UPA (per SPCs):

    1. CYP3A4 inducers (rifampin, barbiturates, carbamazepine, bosentan, felbamate, griseofulvin, oxcarbazepine, phenytoin, St John's Wort, topiramate),
    2. Other hormonal contraceptives including emergency contraception.
21. Use of any medications that can interfere with the metabolism of hormone contraceptives, antibiotics that can interfere with metabolism of hormone contraceptives, and any drugs designated by the FDA as Pregnancy Category D or X.
22. Current participation in any other trial of an investigational medicine or device or participation in the past three months before start of first treatment phase.
23. Headaches with focal neurological symptoms only.
24. Have diastolic blood pressure (BP) >95 mm Hg and systolic BP >145 mm Hg after 5 minutes in sitting position.

    1. Hypertensive subjects who are treatment controlled and in the judgment of the investigator are a good candidate require a waiver for participation.
25. BMI ≥40 kg/m² or having previously undergone bariatric surgery.
26. Have issues or concerns (in the judgment of the investigator) that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study.

    -

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Ovulation inhibition | Approximately 6.5 months
  * Two consecutive serum progesterone values ≥10nMol/L (3ng/mL) within a four day window;
  * A follicle ≥13 mm followed by a single serum progesterone value ≥10nMol/L (3ng/mL) without a second high progesterone level but with follicle disappearance, suggestive of follicular rupture.

SECONDARY OUTCOMES:
Bleeding profile | Approximately 6.5 months
  Total number of bleeding and spotting days per 28 day and 84 day interval, menses duration and intensity, bleeding-related AEs, hematocrit levels, subject's acceptability of treatment.
Follicle growth and rupture | Approximately 6.5 months
  Follicle growth (≥13 mm and ≥15 mm) and rupture assessed using transvaginal ultrasound (TVUS) twice weekly during the 84 day treatment.
Endometrial safety | Approximately 6.5 months
  1. Endometrial thickness by TVUS
  2. Endometrial biopsies during the Baseline cycle at Visit BL2 (Proliferative phase), on Treatment at Visit 22 ± 1 visit (between days 70 -80) OR 7-10 days following any suspected ovulation that occurs after the first 28 days of treatment, and at the end of the recovery period after two full washout cycles during day 7 following start of second menses (Proliferative phase).
Overall subject satisfaction and safety | Approximately 6.5 months

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - California Family Health Council, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado - Denver Anschutz Medical Campus, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - NYU School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati-Holmes Hospital, Cincinnati, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Eastern Virgina Medical School, Norfolk, Virginia